CLINICAL TRIAL: NCT00507832
Title: Evaluation of the Antipruritic Effect of Elidel (Pimecrolimus) in Non-atopic Pruritic Disease
Acronym: CASM981CDE21
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: University Hospital Münster, University Hospital Münster
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SST-Pr-2-2005
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2009-02

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo nodularis
MeSH Terms: interventions — pimecrolimus; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Interindividual design:
  active and comparator (one side each) applied twice daily
  Interventions: Drug: Pimecrolimus
- II Hydrocortisone (Active Comparator): Hydrocortisone, twice daily
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Pimecrolimus — twice daily topical
  Other Names: Elidel Cream 1%
  Arms: I
Drug: Hydrocortisone — twice daily topical
  Other Names: Hydrocortisone HExal
  Arms: II Hydrocortisone
Drug: Pimecrolimus — topical application as a cream twice daily
  Other Names: Elidel 1% Cream
  Arms: I

SUMMARY:
The development of the topical calcineurin inhibitor pimecrolimus resulted in a significant improvement in the treatment of atopic dermatitis. In addition, an excellent amelioration of pruritus could be regularly observed. Up to now, several itchy dermatoses such as chronic irritative hand dermatitis, rosacea, graft-versus-host-disease, lichen sclerosus, prurigo simplex, scrotal eczema, and inverse psoriasis were reported as single cases also to respond to a pimecrolimus treatment.

In prurigo nodularis, pruritus is the main symptom and it is of immediate importance to find an effective antipruritic therapy. Pruritus is regularly severe and therapy refractory to topical steroids or systemic antihistamines. Capsaicin cream is one effective possibility to reduce the itch in these diseases. However, it has to be applied 3 to 6 times daily, rubs off on the clothing and induces burning in erosions. In addition, since no commercial preparation is available, it has to be prescribed in several concentrations. The application of pimecrolimus seems to be promising since it has to be applied twice daily only. Especially in prurigo nodularis we expect a good response as we could demonstrate in single patients. Furthermore it has been published recently that Tacrolimus, another calcineurin inhibitor has been successfully used in the treatment of six patients with prurigo nodularis.

This study is designed to compare the efficacy and safety of pimecrolimus 1% cream and hydrocortisone 1% cream in prurigo nodularis and to investigate the mode of action of the antipruritic effect of the drugs.

DETAILED DESCRIPTION:
Patients will be treated with pimecrolimus cream 1% and hydrocortisone cream 1% twice daily for 8 weeks on diseased skin in a double-blind, randomized within patient comparison (left arm pimecrolimus, right arm hydrocortisone or vice versa). Patients will then enter a 4-week treatment free follow-up period. The overall study duration is 12 months.

The study population will consist of a representative group of 30 adult patients (18 - 70 years of age) with prurigo nodularis from one center in Germany.

Inclusion criteria

* Age: 18 - 70 years
* Diagnosis: Prurigo nodularis
* Pruritus intensity above VAS 3 (Visual analogue scale 0 to 10)
* Nodules on arms and legs (target areas: arms)
* No effective current external or internal antipruritic medication
* Signed informed consent

Exclusion criteria

* prurigo nodularis with massive excoriations and/or local infections
* atopic dermatitis, predisposition for atopic dermatitis
* Itch intensity below VAS 4 (visual analoge scale 0 to 10)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG test. Pregnancy should be ruled out before stating the study by a b-subunit HCG test.
* Females of childbearing potential and not practicing a medically approved, highly effective (low failure rate) method of contraception during and up to at least 4 weeks after the end of treatment. 'Medically approved' contraception may include implants, injectables, combined oral contraceptives, some IUDs (e.g. intrauterine device), sexual abstinence or if the woman has a vasectomized partner.
* active psychosomatic and psychiatric diseases
* History of active malignancy of any organ system
* actual diseases which need therapy and may induce pruritus (e.g. deficiency of iron, zinc)
* Systemic immunosuppression
* Topical use of tacrolimus, pimecrolimus, steroids or capsaicin within 2 weeks prior to study entry
* current and past (within 2 weeks prior to study entry) systemic use of antihistamines, steroids, cyclosporin A and other immunosuppressants, paroxetin, fluvoxamine (selective serotonin reuptake- inhibitors, study possible in case of medication since 6 months due to depression without having any Antipruritic effect) naltrexone and UV-therapy.
* wound healing disturbances, disposition for keloids, current medication which leads to increased bleeding during procedure e.g. acetylsalicylic acid (ASS), marcumar (no suction blister possible)
* History of hypersensitivity to pimecrolimus 1% cream or hydrocortisone 1% cream
* Participation in other clinical studies within the last 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 70 years
* Diagnosis: Prurigo nodularis
* Pruritus intensity above VAS 3 (Visual analoge scale 0 to 10)
* Nodules on arms and legs (target areas: arms)
* No effective current external or internal antipruritic medication
* Signed informed consent

Exclusion Criteria:

* prurigo nodularis with massive excoriations and/or local infections
* atopic dermatitis, predisposition for atopic dermatitis
* Itch intensity below VAS 4 (visual analoge scale 0 to 10)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG test. Pregnancy should be ruled out before stating the study by a b-subunit HCG test.
* Females of childbearing potential and not practicing a medically approved, highly effective (low failure rate) method of contraception during and up to at least 4 weeks after the end of treatment. 'Medically approved' contraception may include implants, injectables, combined oral contraceptives, some IUDs (e.g. intrauterine device), sexual abstinence or if the woman has a vasectomized partner.
* active psychosomatic and psychiatric diseases
* History of active malignancy of any organ system
* actual diseases which need therapy and may induce pruritus (e.g. deficiency of iron, zinc)
* Systemic immunosuppression
* Topical use of tacrolimus, pimecrolimus, steroids or capsaicin within 2 weeks prior to study entry
* current and past (within 2 weeks prior to study entry) systemic use of antihistamines, steroids, cyclosporin A and other immunosuppressants, paroxetin, fluvoxamine (selective serotonin reuptake- inhibitors, study possible in case of medication since 6 months due to depression without having any Antipruritic effect) naltrexone and UV-therapy.
* wound healing disturbances, disposition for keloids, current medication which leads to increased bleeding during procedure e.g. acetylsalicylic acid (ASS), marcumar (no suction blister possible)
* History of hypersensitivity to pimecrolimus 1% cream or hydrocortisone 1% cream
* Participation in other clinical studies within the last 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Hypothesis: pimecrolimus is superior in the reduction of the itch intensity on a visual analogue scale (VAS) compared to hydrocortisone cream 1%. H1: mean value VAS pimecrolimus < mean value VAS hydrocortisone | 12 months

SECONDARY OUTCOMES:
Improvement of total symptom score (papule, nodules, excoriations, crusting, erythema) scored from 0-3 for each single symptom | 12 months
Change of skin neuropeptide content in suction blisters | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Luger, MD, Principal Investigator — Department of Dermatology, University of Münster, Von-Esmarch-Str. 58, D-48149 Münster, Germany
Locations (1):
- Department of Dermtology, University of Münster, Münster, Germany

REFERENCES:
- [Background] Stander S, Stander H, Seeliger S, Luger TA, Steinhoff M. Topical pimecrolimus and tacrolimus transiently induce neuropeptide release and mast cell degranulation in murine skin. Br J Dermatol. 2007 May;156(5):1020-6. doi: 10.1111/j.1365-2133.2007.07813.x. Epub 2007 Mar 28. PMID 17388925
- [Background] Stander S, Luger TA. [Antipruritic effects of pimecrolimus and tacrolimus]. Hautarzt. 2003 May;54(5):413-7. doi: 10.1007/s00105-003-0521-6. Epub 2003 Mar 21. German. PMID 12719860
- [Background] Senba E, Katanosaka K, Yajima H, Mizumura K. The immunosuppressant FK506 activates capsaicin- and bradykinin-sensitive DRG neurons and cutaneous C-fibers. Neurosci Res. 2004 Nov;50(3):257-62. doi: 10.1016/j.neures.2004.07.005. PMID 15488288